CLINICAL TRIAL: NCT03067896
Title: Effect of Adding Dexmedetomidine Versus Magnesium Sulphate to Intrathecal Bupivacaine on Spinal Block and Neonatal Outcome in Uncomplicated Caesarean Delivery
Brief Title: Dexmedetomidine Versus Magnesium Sulphate for Caesarean Delivery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed talaat ahmed aly, Assisstant lecturer of anesthesia and intensive care, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: assuit university
Record Dates: First submitted 2015-07-12; First posted 2017-03-01 (Actual); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Cesarean Section
Keywords: spinal block; stress response; dexmedetomidine; intrathecally
MeSH Terms: conditions — Fractures, Stress | interventions — Bupivacaine; Dexmedetomidine; Magnesium Sulfate

ARMS (3):
- Group C (Active Comparator): Patients will receive intrathecal hyperbaric bupivacaine 12.5 mg in 2.5 ml
  Interventions: Drug: Bupivacaine
- Group D (Active Comparator): Patients will receive intrathecal hyperbaric bupivacaine 10 mg in 2 ml with dexmdetomidine 5 µg in 0.5 ml normal saline .
  Interventions: Drug: Dexmedetomidine
- Group M (Active Comparator): Patients will receive intrathecal hyperbaric bupivacaine 10 mg in 2 ml with magnesium sulfate 50 mg in 0.5 ml normal saline .
  Interventions: Drug: Magnesium Sulfate

INTERVENTIONS:
Drug: Bupivacaine — Patients will receive intrathecal hyperbaric bupivacaine 12.5 mg in 2.5 ml
  Arms: Group C
Drug: Dexmedetomidine — Patients will receive intrathecal hyperbaric bupivacaine 10 mg in 2 ml with dexmdetomidine 5 µg in 0.5 ml normal saline
  Arms: Group D
Drug: Magnesium Sulfate — Patients will receive intrathecal hyperbaric bupivacaine 10 mg in 2 ml magnesium sulfate 50 mg in 0.5 ml normal saline
  Arms: Group M

SUMMARY:
Regional anesthesia has become more popular in cesarean deliveries because most of the parturients prefer being awake during the birth process. In addition, regional anesthesia may be a safer method than general. In spinal anesthesia local anesthetics alone may not be enough for an effective postoperative analgesia and hemodynamic stability of the patient wich is crucial during cesarean section. So far many adjuvants have been used to augment the analgesia produced by intrathecal local anesthetics and to reduce their adverse effects .

Various intrathecal adjuvants to local anaesthetics have found to improve the quality and extend duration of spinal block. Prolongation of duration of spinal block is desirable both for long procedures and for postoperative pain relief. Efficacy and safty of intrathecal magnesium as analgesic adjuvant has been tested by several clinical trails in recent years.Antinociceptive effect of magnesium appears to be relevant for the management of chronic and post operative pain. These effects are primarily based on regulation of calcium influx in to the cell. Magnesium blocks calcium influx and non competitively antagonizes NMDA channels. NMDA receptor signelling plays an impartent in determining the duration of acute pain3).) addition of magnesium to spinal anaesthesia improved postoperative analgesia in orthopedic setting. addition of intrathecal magnesium sulfate to 10 mg bupivacaine plus 25µg fentanyl prolonged spinal anaesthesia in patients undergoing lower extremity surgery.

Dexmedetomidine is a highly selective 2-adrenergic agonist which has been used as pre-medication and as an adjuvant to general anesthesia.Dexmedetomidine have several beneficial actions during perioperative period. They decrease sympathetic tone with attenuation of the neuroendocrine and haemodynamic response to anaesthesia and surgery, reduce anaesthetic and opiod requirement, cause sedation and analgesia. Dexmedetomidine was first introduced into clinical practice as a short term intravenous sedative in intensive care. Like any other adjuvant dexmedetomidine is not free from adverse effects. Use of dexmedetomidine is often associated with a decrease in heart rate and blood pressure.Dexmedetomidine was used to enhance the analgesic property of local anaesthetics like lidocaine bupivacaine and ropivacaine. In vivo and in vitro studies indicated that these local anaesthetics had significant neurotoxicity. Dexmedetomidine showed protective or growth promoting properties in tissues, including nerve cells from cortex. Intrathecal dexmedetomidine has a neuroprotective effect similar to methylprednisolone.

The mechanism by which intrathecal alpha 2-adrenergic agonists prolong the motor and sensory block of local anesthetics is not clear. It may be an additive or synergistic effect secondary to the different mechanisms of action of local anesthetic and alpha 2 adrenergic agonist. The local anesthetics act by blocking sodium channels, whereas the alpha 2 adrenergic agonist acts by binding to pre synapyic C fibre and post synaptic dorsal horn neurons. Intrathecal alpha 2 adrenergic agonist produce analgesia by depressing the realease of C fibre transmission by hyperpolarization of post synaptic dorsal horn neurons. Li et al observed that Glutamate is involved in excitatory neurotransmission nociception and plays an essential role in relaying noxious stimuli in the spinal cord. Intrathecal injection of alpha 2 adrenergic agonists produces potent antinociceptive effects by altering spinal neurotransmitter release and effectively treats acute pain.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 45 years
2. Undergo elective cesarean section under spinal anesthesia.
3. ASA physical status Ӏ-ӀӀ .
4. Singleton pregnancy .
5. At least 36 weaks gestation .

Exclusion Criteria:

1. Women with a history of cardiac , liver , or kidney diseases .
2. Women with allergy to amide local anesthetics or medications included in the study .
3. Women with any neurological problem .
4. Any contraindication of regional anesthesia .
5. Women with evidence of intrauterine growth restriction or fetal compromise .
6. Failed or insatisfactory spinal block .

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2015-06; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale | 6 hours
  analgesia will be given if VAS is 4 or more

SECONDARY OUTCOMES:
heart rate | 6 hours
  effect of study drugs on the maternal heart rate
blood pressure | 6 hours
  effect of study drugs on the maternal mean blood pressure

OTHER OUTCOMES:
APGAR Score | 5 minutes
  effect of study drugs on the APGAR fetal outcome
plasma concentration of stress hormones | 3 hours
  effect of study drugs on the stress hormones levels

CONTACTS AND LOCATIONS:
Overall Officials: Zain E. Hassan, MD, Study Director — Assiut University
Locations (1):
- Ahmed Talaat Ahmed, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mostafa MF, Herdan R, Fathy GM, Hassan ZEAZ, Galal H, Talaat A, Ibrahim AK. Intrathecal dexmedetomidine versus magnesium sulphate for postoperative analgesia and stress response after caesarean delivery; randomized controlled double-blind study. Eur J Pain. 2020 Jan;24(1):182-191. doi: 10.1002/ejp.1476. Epub 2019 Sep 12. PMID 31461801